CLINICAL TRIAL: NCT03691922
Title: Randomized Control Trial of Ultrasound-Guided Erector Spinae Block Versus Shoulder Periarticular Anesthetic Infiltration for Pain Control After Arthroscopic Shoulder Surgery
Brief Title: Erector Spinae Block Versus Shoulder Periarticular Anesthetic Infiltration for Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 4668
Record Dates: First submitted 2018-09-18; First posted 2018-10-02 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-08

CONDITIONS: Arthroscopic Shoulder Surgery
Keywords: Shoulder; Pain; Erector Spinae Plane block; Surgery; Arthroscopy; Periarticular infiltration; Post-Anesthesia Care Unit; Day Surgery Unit; Regional anesthesia; Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Parapsychology; Dental Occlusion; Bupivacaine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Block (Active Comparator): Preoperative US guided active Erector Spinae Plane (ESP) block and a saline PAI
  Interventions: Procedure: Erector Spinae Plane (ESP) Block
- PAI with LA (Other): Preoperative US guided ESP blockade with saline and an active Periarticular Infiltration (PAI)
  Interventions: Procedure: Periarticular Infiltration (PAI)

INTERVENTIONS:
Procedure: Erector Spinae Plane (ESP) Block — 1. Preoperative US guided ESP blockade using 30 mL of 0.25% bupivacaine with 5 mcg/mL of epinephrine, injected in 5-mL aliquots through the needle (maximum of 3 mg/kg)
  2. PAI of 30 mL of saline at the end of the surgical procedure on the operated side rotator cuff, injected in 5-mL aliquots through the needle
  Other Names: 0.25% bupivacaine with 5 mcg/mL of epinephrine & PAI with 30 mL of saline
  Arms: ESP Block
Procedure: Periarticular Infiltration (PAI) — 1. Preoperative US guided ESP blockade using 30 mL of saline, injected in 5-mL aliquots through the needle
  2. PAI of 30 mL of 0.25% bupivacaine with 5 mcg/mL of epinephrine at the end of the surgical procedure on the operated side rotator cuff, injected in 5-mL aliquots through the needle
  Other Names: ESP block with 30 mL of saline & PAI with 30 mL of 0.25% bupivacaine with 5 mcg/mL of epinephrine
  Arms: PAI with LA

SUMMARY:
Arthroscopic shoulder surgery is a common and minimally invasive procedure utilized for different shoulder pathologies, but it is often associated with moderate to severe postoperative pain that may interfere with patients' well-being and course of recovery. By using an effective analgesic technique with few side effects, a patient may experience less pain after surgery, have a shortened hospital stay, and endure less nausea, vomiting, or excessive drowsiness that are associated with the use of opioids to manage postoperative pain. Periarticular infiltration (PAI) with local anesthetic (LA) has been used for shoulder surgery pain management, but the more effective interscalene nerve block (ISNB) is the current gold standard analgesic modality despite risk of significant side effects including diaphragm paralysis and rebound pain. In this study, the investigators want to look at the effectiveness and safety profile of a novel technique for pain management after shoulder surgery that has the potential to provide successful pain relief with minimal risk of side effects. Half of the patients will be randomly selected to receive the novel nerve block called the Erector Spinae Plane (ESP) block while the other half will receive a more standard PAI of local anesthetic to numb the shoulder. Patients' pain intensity and opioid consumption in the post-anesthesia care unit (PACU) as well as during the first 24 hours after surgery will be evaluated. Any complications from the interventions will also be noted. The investigators predict that the ESP block will provide superior analgesia compared to PAI for these shoulder arthroscopy patients.

DETAILED DESCRIPTION:
The use of opioids to manage immediate postoperative pain is frequently associated with nausea, vomiting, respiratory depression, hormonal effects and dysphoria. As such, achieving pain control while minimizing opioid use is critical, since more than 60% of unplanned prolonged hospitalizations and hospital readmissions are thought to be related to inadequate pain control or to side effects of opioids. A number of techniques have been used to achieve good pain control after arthroscopic shoulder surgery, including periarticular infiltration (PAI) with local anesthetic (LA) and regional anesthetic nerve blocks. Although PAI in the shoulder has been shown to decrease shoulder pain and opioid consumption, it is not as effective as regional blocks such as the interscalene nerve block (ISNB), which is the current gold standard. Nevertheless, the ISNB is potentially associated with significant side effects including persistent neurologic complications, rebound pain, phrenic nerve palsy, respiratory distress, cardiac arrest pneumothorax and central nerve toxicity. In view of this, investigating alternate regional blocks having the potential for good pain relief with minimal side effects is important. The Erector Spinae Plane (ESP) block can be considered as a modification of thoracic paravertebral block (PVB) that blocks thoracic spinal nerves using injections outside of the conventional paravertebral space. It is performed under ultrasound (US) by injecting local anesthetic deep to the erector spinae muscle at the interfascial space between either the erector spinae muscle and the rhomboid major muscle (higher up), or between the erector spinae muscle and the external intercostal muscles, at lower sites. Cadaveric studies of ultrasound-guided ESP blocks with methylene blue dye and subsequent dissection, as well an ESP block with a dye mixture and CT scanning demonstrated that when injecting deep into the erector spinae, the block likely affects the ventral and dorsal rami leading to the sensory blockade. The advantages include its simplicity and safety by limiting the risk of nerve damage and pneumothorax. Various case reports have demonstrated the ESP block to be successful for abdominal, breast and axillary, and other surgery types, and a recent case report described the successful management of chronic shoulder pain without motor blockade, with ESP performed at T3 level. The investigators conducted a systematic review via Pubmed to identify studies that have utilized ESP for post-surgical shoulder pain. Out of 77 reports, the investigators did not identify any comparative studies looking at the potential of ESP for shoulder surgery pain. The investigators also looked into ongoing and proposed trials of ESP by looking into clinicaltrials.gov. The investigators identified 21 studies including some randomized controlled trials (RCT) for thoracic surgery and general surgery population, but none for shoulder surgeries. Given the importance of providing adequate analgesia for arthroscopic shoulder surgery and lack of consensus amongst surgeons and anesthesiologists for the optimal analgesic technique, this trial will help establish the effectiveness of the ESP block in pain control after shoulder arthroscopy and define its safety profile. The results of this trial will allow the clinician to inform patients accurately regarding the benefits and risks of the block and thus guide the clinical practice of this block for shoulder arthroscopy. If proven to be effective, it may be used as an alternative to ISNB, especially in cases where ISNB is contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* elective arthroscopic shoulder joint surgeries admitted for day surgical procedure
* an ability to provide informed consent

Exclusion Criteria:

* not willing
* contraindications to spinal injections as per the American Society of Regional Anesthesia and Pain (ASRA) guidelines
* known allergy to LA
* allergy to all opioid medications
* diagnostic shoulder arthroscopic procedures
* inability to understand or comprehend in English language
* history of daily opioid medication use for the last one month
* patients with planned overnight hospital stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-07-06 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Recovery room resting pain score | At 30 minutes post-admission to recovery room
  Using the patient-reported numeric rating scale (0-10) (0 is no pain and 10 is worst pain imaginable).

SECONDARY OUTCOMES:
Day Surgery Unit resting pain score | At 5 hours post-operatively
  Using the patient-reported numeric rating scale (0-10) (0 is no pain and 10 is worst pain imaginable).
Pain scores with movement | At 30 minutes post-admission to recovery room and 5 hours post-operatively
  Using the patient-reported numeric rating scale (0-10). (0 is no pain and 10 is worst pain imaginable). Participants will be asked to sit up from lying down position.
Opioid usage | At 2 hours post-operatively and 5 hours post-operatively
  All opioids administered in recovery room and day surgery unit will be converted into Morphine Equivalent Units per patient according to accepted standards.
Incidence of moderate to severe postoperative nausea-vomiting | At 2 hours post-operatively and 5 hours post-operatively
  Using a 0-3 scale (0 is none and 3 severe nausea-vomiting)
Incidence of moderate to severe itching | At 2 hours post-operatively and 5 hours post-operatively
  Using a 0-3 scale (0 is none and 3 severe itching)
Incidence of ipsilateral diaphragmatic paralysis | 30 minutes post-admission to recovery room
  Diagnosed based on the findings in an anterior posterior chest using ultrasound , with the criteria of "a right hemidiaphragm sitting >2 cm higher than its left counterpart or a left hemidiaphragm sitting equal or higher than the right hemidiaphragm".
Incidence of respiratory depression | At 2 hours post-operatively and 5 hours post-operatively
  Opioids discontinued by the Acute Pain Service or recovery room nursing due to concerns of respiratory depression by nursing staff.
Incidence of local anesthetic toxicity | At 2 hours post-operatively and 5 hours post-operatively
  Based on clinical symptoms and signs of local anesthetic toxicity as diagnosed by the attending physician.
Sensory blockade | At 30 minutes post-admission to recovery room
  Seven sensory dermatomes corresponding to shoulder and upper arm and their blockade to cold sensation will be noted. The extent of blockade between the two groups will be compared by their median and range.
Patient Satisfaction with Postoperative Analgesia | At 5 hours post-operatively and 24 hours post-operatively
  Using a 7-item Likert scale (1 is extremely satisfied and 7 is extremely dissatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Shanthanna, MD, Principal Investigator — St. Joseph's Healthcare Hamilton/McMaster University; Bashar Alolabi, MD, Principal Investigator — St. Joseph's Healthcare Hamilton; Mark Czuczman, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Fontana C, Di Donato A, Di Giacomo G, Costantini A, De Vita A, Lancia F, Caricati A. Postoperative analgesia for arthroscopic shoulder surgery: a prospective randomized controlled study of intraarticular, subacromial injection, interscalenic brachial plexus block and intraarticular plus subacromial injection efficacy. Eur J Anaesthesiol. 2009 Aug;26(8):689-93. doi: 10.1097/eja.0b013e32832d673e. PMID 19593887
- [Background] Manchikanti L, Fellows B, Ailinani H, Pampati V. Therapeutic use, abuse, and nonmedical use of opioids: a ten-year perspective. Pain Physician. 2010 Sep-Oct;13(5):401-35. PMID 20859312
- [Background] Chung F, Ritchie E, Su J. Postoperative pain in ambulatory surgery. Anesth Analg. 1997 Oct;85(4):808-16. doi: 10.1097/00000539-199710000-00017. PMID 9322460
- [Background] Barber FA, Herbert MA. The effectiveness of an anesthetic continuous-infusion device on postoperative pain control. Arthroscopy. 2002 Jan;18(1):76-81. doi: 10.1053/jars.2002.25976. PMID 11774146
- [Background] Merivirta R, Kuusniemi KS, Aantaa R, Hurme SA, Aarimaa V, Leino KA. The analgesic effect of continuous subacromial bupivacaine infusion after arthroscopic shoulder surgery: a randomized controlled trial. Acta Anaesthesiol Scand. 2012 Feb;56(2):210-6. doi: 10.1111/j.1399-6576.2011.02606.x. PMID 22236345
- [Background] Harvey GP, Chelly JE, AlSamsam T, Coupe K. Patient-controlled ropivacaine analgesia after arthroscopic subacromial decompression. Arthroscopy. 2004 May;20(5):451-5. doi: 10.1016/j.arthro.2004.03.004. PMID 15122133
- [Background] Warrender WJ, Syed UAM, Hammoud S, Emper W, Ciccotti MG, Abboud JA, Freedman KB. Pain Management After Outpatient Shoulder Arthroscopy: A Systematic Review of Randomized Controlled Trials. Am J Sports Med. 2017 Jun;45(7):1676-1686. doi: 10.1177/0363546516667906. Epub 2016 Oct 13. PMID 27729319
- [Background] Uquillas CA, Capogna BM, Rossy WH, Mahure SA, Rokito AS. Postoperative pain control after arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2016 Jul;25(7):1204-13. doi: 10.1016/j.jse.2016.01.026. Epub 2016 Apr 11. PMID 27079219
- [Background] Shin SW, Byeon GJ, Yoon JU, Ok YM, Baek SH, Kim KH, Lee SJ. Effective analgesia with ultrasound-guided interscalene brachial plexus block for postoperative pain control after arthroscopic rotator cuff repair. J Anesth. 2014 Feb;28(1):64-9. doi: 10.1007/s00540-013-1681-x. Epub 2013 Aug 1. PMID 23903900
- [Background] Misamore G, Webb B, McMurray S, Sallay P. A prospective analysis of interscalene brachial plexus blocks performed under general anesthesia. J Shoulder Elbow Surg. 2011 Mar;20(2):308-14. doi: 10.1016/j.jse.2010.04.043. Epub 2010 Aug 13. PMID 20708419
- [Background] Webb BG, Sallay PI, McMurray SD, Misamore GW. Comparison of Interscalene Brachial Plexus Block Performed With and Without Steroids. Orthopedics. 2016 Nov 1;39(6):e1100-e1103. doi: 10.3928/01477447-20160819-02. Epub 2016 Aug 30. PMID 27575034
- [Background] Candido KD, Sukhani R, Doty R Jr, Nader A, Kendall MC, Yaghmour E, Kataria TC, McCarthy R. Neurologic sequelae after interscalene brachial plexus block for shoulder/upper arm surgery: the association of patient, anesthetic, and surgical factors to the incidence and clinical course. Anesth Analg. 2005 May;100(5):1489-1495. doi: 10.1213/01.ANE.0000148696.11814.9F. PMID 15845712
- [Background] Nam YS, Jeong JJ, Han SH, Park SE, Lee SM, Kwon MJ, Ji JH, Kim KS. An anatomic and clinical study of the suprascapular and axillary nerve blocks for shoulder arthroscopy. J Shoulder Elbow Surg. 2011 Oct;20(7):1061-8. doi: 10.1016/j.jse.2011.04.022. Epub 2011 Aug 11. PMID 21839653
- [Background] Costache I, de Neumann L, Ramnanan CJ, Goodwin SL, Pawa A, Abdallah FW, McCartney CJL. The mid-point transverse process to pleura (MTP) block: a new end-point for thoracic paravertebral block. Anaesthesia. 2017 Oct;72(10):1230-1236. doi: 10.1111/anae.14004. Epub 2017 Aug 1. PMID 28762464
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Hamilton DL, Manickam B. The Erector Spinae Plane Block. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):276. doi: 10.1097/AAP.0000000000000565. No abstract available. PMID 28207652
- [Background] Forero M, Rajarathinam M, Adhikary SD, Chin KJ. Erector spinae plane block for the management of chronic shoulder pain: a case report. Can J Anaesth. 2018 Mar;65(3):288-293. doi: 10.1007/s12630-017-1010-1. Epub 2017 Nov 13. PMID 29134518
- [Background] Tran DQ, Elgueta MF, Aliste J, Finlayson RJ. Diaphragm-Sparing Nerve Blocks for Shoulder Surgery. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):32-38. doi: 10.1097/AAP.0000000000000529. PMID 27941477
- [Background] Abdallah FW, Halpern SH, Aoyama K, Brull R. Will the Real Benefits of Single-Shot Interscalene Block Please Stand Up? A Systematic Review and Meta-Analysis. Anesth Analg. 2015 May;120(5):1114-1129. doi: 10.1213/ANE.0000000000000688. PMID 25822923
- [Derived] Czuczman M, Shanthanna H, Alolabi B, Moisiuk P, O'Hare T, Khan M, Forero M, Davis K, Moro J, Vanniyasingam T, Thabane L. Randomized control trial of ultrasound-guided erector spinae block versus shoulder periarticular anesthetic infiltration for pain control after arthroscopic shoulder surgery: Study protocol clinical trial (SPIRIT compliant). Medicine (Baltimore). 2020 Apr;99(15):e19721. doi: 10.1097/MD.0000000000019721. PMID 32282729